CLINICAL TRIAL: NCT00532870
Title: Laparoscopic Intraperitoneal Mesh Repair of Ventral Hernia: Comparison to Conventional Mesh Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mfms1861964
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Hernia, Ventral
Keywords: laparoscopy; ventral hernia; mesh; Ventral hernias are the second most common type of abdominal hernias after inguinal hernias.; The majority of ventral hernias are incisional hernias that develop in 11% to 20% of patients who undergo Laparotomy .; Surgeons have struggled to reduce the morbidity from incarceration (6% to 15% of cases) and strangulation (2%) of these hernias.
MeSH Terms: conditions — Hernia, Ventral | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): laparoscopy
  Interventions: Other: laparoscopic

INTERVENTIONS:
Other: laparoscopic

SUMMARY:
The laparoscopic repair of ventral hernias is still a controversial therapeutic option. To evaluate the efficacy and safety of laparoscopic repair we compare the results of the open and laparoscopic repair of ventral hernia,. 53 patients were undergo laparoscopic or open repair of ventral hernia . All defects were estimated to be larger than 5 cm in diameter. Twenty six patients underwent attempted laparoscopic ventral hernia repair (LVHR) with mesh and twenty seven patients underwent open ventral hernia repair (OVHR) with mesh

DETAILED DESCRIPTION:
Between March 2003 and December 2004, 53 patients (16 males and 37 females) with ventral hernias were treated by a laparoscopic or open approach. Patients were divided into two groups: one group underwent laparoscopic repair with GORE-TEX Dual Mesh, and the other group underwent open repair with proline mesh. Informed written consents were obtained from all patients.

Inclusion criteria involved any patient aged over 30 years, medical fitness for general anesthesia, the absence of coagulopathy, and hernial defect ≥ 5 cm in any dimension or recurrent hernias. Exclusion criteria were neoplastic patients, immune compromised patients, mentally incompetent patients and those who refused to give signed consents.

Demographic features, operative details and postoperative outcomes were collected prospectively and included patient age, gender, body mass index (BMI) (weight in kg/height in m2), number of prior abdominal operations, number of previous hernia repairs, technique of repair, size of facial defect, type of prosthetic mesh, operating time, conversion rate, length of hospital stay, operative and postoperative complications, and hernia recurrences.

Thirty-seven patients presented with an incisional hernia (12 upper midline, 15 lower midline, and 10 transverse abdominal), 8 had an epigastric hernia, 8 had an periumbilical hernia, . All defects were estimated to be larger than 5 cm in diameter.

Standard bowel preparation was undertaken for every patient on the day before the operation. Prophylactic short-term antibiotic therapy with a one gram of third-generation cephalosporin was also administered routinely two hours before the operation. Nasogastric suction and bladder catheterization were used routinely during the operation only. All operations were performed under general anesthesia; Open mesh repair was done as described else where (9, 10).

Operative Procedure of laparoscopic ventral hernia repair:

pneumoperitoneum was established by using a Verses needle. The initial entry site was usually just inferior to the tip of the eleventh rib to establish a 15 mmHg pneumoperitoneum for exploration of the abdomen. One 10-mm trocar and three to five 5-mm trocars were then placed outside the perimeter of the hernia. Adhesiolysis was performed to free the anterior abdominal wall and identify the hernia defect. The peritoneal sac was not reduced and the mesh was placed in an intraabdominal position.

The mesh was prepared to extend 3 to 5 cm beyond the hernia defect. Four anchoring sutures were placed in the corners of the mesh, which was then introduced into the abdomen via a 10-mm port. The sutures were secured across the full thickness of the abdominal wall with the use of a laparoscopic suture passer. A laparoscopic mesh stapler device was used to place 5-mm spiral staples at 1-cm intervals around the mesh edge. . No drains were placed.

Postoperative management intravenous analgesia was administered postoperatively. All patients were encouraged to move as soon as possible. Postoperatively, the severity of pain was assessed daily by a visual analogue scale (VAS) on a scale from 0 (no pain) to 10 (worst pain). Upon discharge, all patients were taught to complete a pain score chart at home for daily documentation of pain score at rest and on coughing.

Follow up at the surgical Clinic was scheduled at 1 week, 8 weeks and 1 and 2 years after operation for assessment of postoperative complications: seromas (collection of fluid persisting > 4 weeks or causing local discomfort), hematomas, infection, abdominal wall pain, bowel obstruction, recurrences, aesthetic evaluation. The pain score charts were collected by the surgeon at the surgical clinic. All complications were recorded and clinical recurrence was documented during follow up.

Also, the outcome evaluation was measured by the duration of return to activity, pain free return to activity, return to work and pain free return to work.

Statistical analysis Variables measured on a nominal scale were analyzed in the form of 2 x K tables and Fisher's exact test when appropriate. Variables measured on an ordinal scale were analyzed by kruskal Wallis test. All tests were two tailed and made at a level of significance of < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 30 years
* Medical fitness for general anesthesia
* The absence of coagulopathy, and hernial defect ≥ 5 cm in any dimension or recurrent hernias.

Exclusion Criteria:

Exclusion criteria were:

* Neoplastic patients
* Immune compromised patients
* Mentally incompetent patients; and
* Those who refused to give signed consents.

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-03; Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: tarek mahdy, md, Principal Investigator — Mansoura University Hospital
Locations (2):
- Egypt (2):
  - Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Al Mansurah